CLINICAL TRIAL: NCT01764620
Title: Effects of Muscle Fatigue and Scapular Taping on Shoulder Kinematics of Overhead Athletes
Brief Title: Effects of Muscle Fatigue and a Taping Technique on Shoulder Motion of Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Gisele Garcia Zanca, MSc, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 040/2011
Record Dates: First submitted 2012-12-18; First posted 2013-01-09 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Shoulder Injury; Muscle Fatigue
Keywords: shoulder; muscle fatigue; kinematics; athletes
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Other): In this session, the athletes will be evaluated before and after the fatigue protocol, without any taping application.
  Interventions: Other: Fatigue protocol
- Kinesio taping (Experimental): A kinesio taping technique for facilitating lower trapezius muscle function will be applied just before fatigue protocol and removed after in the end of the evaluation session.
  Interventions: Other: Elastic taping applied with tension; Other: Fatigue protocol
- Sham (Sham Comparator): A similar technique, using the same tape, will be applied but without any tension (tension is considered to be the therapeutic effect). The tape will be applied just before the fatigue protocol and removed in the end of the session.
  Interventions: Other: Elastic taping applied without tension; Other: Fatigue protocol

INTERVENTIONS:
Other: Elastic taping applied with tension
  Arms: Kinesio taping
Other: Elastic taping applied without tension
  Arms: Sham
Other: Fatigue protocol

SUMMARY:
The purpose of this study is to investigate the effects of muscle fatigue in the scapular kinematics of overhead athletes with and without using a kinesio taping technique for facilitating lower trapezius function. The hypothesis is that the taping technique could compensate for the negative effects caused by muscle fatigue in the scapular kinematics of healthy overhead athletes.

DETAILED DESCRIPTION:
Muscle fatigue is a potential cause of shoulder injuries in overhead athletes. Considering the important role of lower trapezius for functional scapular stability, it is suggested that a kinesio taping technique for facilitating its function could compensate for the negative effects of muscle fatigue on scapular kinematics. This is a randomized crossover study and all included athletes will be evaluated in three sessions, with a period of seven days between them: Control (fatigue protocol, without taping), Kinesio Taping (fatigue protocol with elastic taping applied with tension) and Sham (fatigue protocol with taping applied without tension). During each session, tridimensional kinematics of scapula and humerus and electromyography of serratus anterior and trapezius (upper and lower portions) muscles of dominant shoulder will be evaluated, during scaption and throwing movements, immediately before and immediately after the fatigue protocol.The changes in scapular movements (before versus after the fatigue protocol) will be compared among the sessions.

ELIGIBILITY:
Inclusion Criteria:

* Overhead athletes regularly training;
* No report of shoulder pain in the last 6 months.

Exclusion criteria:

* Previous shoulder or neck surgery;
* Previous shoulder dislocation.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-12 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Changes in scapular internal/external rotations, upward/downward rotations and anterior/posterior tilt movements | An average of 3 minutes before and an average of 3 minutes after the fatigue protocol, in each of the 3 evaluation sessions.
  Scapular 3D kinematics will be measured during arm elevation and throwing movements, in two moments (an average of 3 minutes before and an average of 3 minutes after the fatigue protocol) in each one of the 3 sessions. The evaluation session will have and interval of 7 days between them, and in each one the athletes will perform the fatigue protocol using either a kinesio taping application, or a sham application or without using any taping, in random order. The changes in each session (before and after fatigue) will be compared among the sessions (without taping, with kinesio taping application and sham application).

SECONDARY OUTCOMES:
Changes in the median frequency of electromyographic signal from upper and lower trapezius and serratus anterior muscles. | An average of 3 minutes before and an average of 3 minutes after the fatigue protocol, in each of the 3 evaluation sessions.
  Electromyographic median frequency will be measured from upper and lower trapezius and serratus anterior muscles in order to determine muscle fatigue development and if the changes depending on the intervention used. These assessments will be performed in two moments (an average of 3 minutes before and an average of 3 minutes after the fatigue protocol) in each one of the 3 sessions(with an interval of 7 days between them). In each session the athletes will perform the fatigue protocol using either a kinesio taping application, or a sham application or without using any taping, in random order.The changes in each session (before and after fatigue) will be compared among the sessions (without taping, with kinesio taping application and sham).

CONTACTS AND LOCATIONS:
Overall Officials: Gisele G Zanca, MSc, Principal Investigator — Universidade Federal de Sao Carlos; Stela M Mattiello, PhD, Study Director — Universidade Federal de Sao Carlos
Locations (1):
- Universidade Federal de São Carlos, São Carlos, São Paulo, Brazil